CLINICAL TRIAL: NCT07165925
Title: A Gamified Instrumental Musical Training to Enhance Resilience of Underprivileged School-aged Children at Risk of Mental Health Problems: A Randomised Controlled Trial
Brief Title: Musical Training to Enhance Resilience of Underprivileged School-aged Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Tan, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRE-2024.498
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Resilience; Depressive Symptom; Anxiety
Keywords: Musical training; Resilience; underprivileged children; mental health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified musical training (Experimental): Participants in the gamified musical training group will receive weekly 1-hour lessons on a musical instrument for 6 months, delivered by professionally certified musicians. The intervention will be conducted in small groups (7-8 children/group). Two types of musical instruments (keyboard and ukulele) will be assigned to the participants based on their preferences.
  Interventions: Behavioral: Gamified music training
- Active placebo control group (Placebo Comparator): Participants in the active placebo control group will participate in weekly 1-hour group-based (7-8 children/group) indoor community leisure activities for 6 months.
  Interventions: Behavioral: Active placebo intervention

INTERVENTIONS:
Behavioral: Gamified music training — Instrumental musical training will progress from basic (playing simple notes) to advanced levels (playing an entire song). Key training elements will include fundamental music knowledge and skills, music improvisation, rhythm, and pitch identification exercises. In particular, the core concepts of resilience will be incorporated into the training process through various gamified music activities.
  Arms: Gamified musical training
Behavioral: Active placebo intervention — Participants in the active placebo control group will participate in weekly 1-hour group-based indoor community leisure activities for 6 months. These activities will include (i) drawing, (ii) drama workshops, (iii) cartoon film screenings, (iv) handcraft workshops, (v) board games, and (vi) exercise classes. Each activity will span for four sessions, that is, totally 24 sessions and will be delivered by trained staff at the study centres of the collaborating non-governmental organisations.
  Arms: Active placebo control group

SUMMARY:
This is a multi-centre randomised controlled trial aims to examine the effects of a group-based gamified instrumental musical training in enhancing resilience (primary outcome), reducing psychological distress (depressive symptoms and anxiety), enhancing self-esteem, and improving HRQoL (secondary outcomes) among underprivileged school-aged children at risk of mental health problems (depression and anxiety) during a 12-month follow-up.

DETAILED DESCRIPTION:
Background: Child poverty is a prominent global health issue owing to its detrimental impact on a child's physical and psychosocial well-being. Nearly 356 million children lived in extreme poverty globally before the pandemic and this is estimated to worsen significantly. children growing up in poverty are more vulnerable to its effect and have an increased risk of psychosocial and developmental problems than children from affluent families. The impact of poverty is not only immediate during childhood but can persist into adulthood. Previous studies have shown that Chinese children from low-income families reported significantly higher levels of depressive symptoms, lower levels of self-esteem, quality of life, and life satisfaction than children from affluent families.

Therefore, there is an urgent need to design and implement promising and novel approaches for this vulnerable population to prevent children from developing mental health problems.

Growing evidence indicates the importance of fostering children's resilience to enable them to cope with adversity. Research found that resilience exerts a protective effect on the mental well-being of individuals facing adversity (i.e. exposure to poverty).

Emerging evidence reveals the promising effects of musical training of music-based interventions on enhancing resilience and psychosocial outcomes in paediatric populations. Yet, whether music-based interventions can enhance resilience in underprivileged school-aged children remains unclear.

If the proposed instrumental musical training programme is proven to be effective and sustainable, it can be recommended as usual care in the community care service for underprivileged children.

Hypothesis to be tested: Participants who receive the 6-month gamified instrumental musical training would report higher levels of resilience, reduced levels of psychological distress (depressive symptoms and anxiety), higher self-esteem, and better QoL than the placebo control group.

Design and subjects: A mulit-centre assessor-blind, randomised controlled trial will be conducted following the CONSORT guidelines; 174 underprivileged children aged 8 to 12 who are at risk of depression and/or anxiety will be randomised 1:1 to intervention or control groups.

Instruments: Validated questionnaires (RSES, CES-DC, SAS-C, RS10,and PedsQL 4.0).

Interventions: Weekly one-hour group-based gamified instrumental musical training session delivered by certified musicians for 6 months. The control group will receive weekly one-hour group-based indoor community leisure activities for 6 months.

Main outcome measures: Data collection will be conducted at baseline (T0), 6-month (T1;immediately post-intervention), 9-(T2), and 12-month(T3). The primary outcome is resilience level. Secondary outcomes include psychological distress (i.e., depressive symptoms and anxiety levels), self-esteem, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese children aged 8-12 years.
* Able to read Chinese and communicate in Cantonese/Mandarin.
* From low-income families.
* Have a risk of mental health problems, specifically depression and/or anxiety (determined through screening during the recruitment process using the Center for Epidemiological Studies Depression Scale for Children, with a cut-off score of ≥16 indicating a high risk of depression, and/or the State Anxiety Scale for Children, with scores between 36 and 60 indicating a significant level of anxiety)

Exclusion Criteria:

* Have chronic health conditions, cognitive and learning difficulties
* if they or their siblings are currently receiving or have received any music-based interventions before the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Resilience | Change from baseline to 12-month post-intervention
  Children's resilience will be measured by the Resilience Scale for Children- 10 (RS10) which was developed based on the Resilience Scale originally developed by Wagnild and Young. Total scores ranging from 10 to 40, with higher scores indicate higher levels of resilience.

SECONDARY OUTCOMES:
Social competence aspect of resilience | Change from baseline to 12-month post-intervention
  The Chinese version of Child Behaviour Checklist - Parent Report Form (CBCL) will be used as an objective measure in assessing children's social competency aspect of resilience. The CBCL is a 118-item scale for assessing a range of emotional and behavioural problems among school-aged children aged 6 to 18 years old. The 20-item social competence scale of CBCL will be used to assess social competency aspect of resilience of children. These 20 items will focus on children's (i) involvement in activities, (ii) social interaction patterns and (iii) school performance.
Depressive symptoms | Change from baseline to 12-month post-intervention
  The Chinese version of the Center for Epidemiological Studies Depression Scale for Children (CES-DC) will be used to assess the participants' depressive symptoms. It consists of 20 items which are rated on a 4- point Likert scale from 0 to 3 (0= "not at all", 3= "a lot") regarding the children' feelings and experiences of last week. Possible score ranges from 0 to 60, higher scores indicate higher level of depression. The cut-off score of this scale is 16, indicating the children are currently experiencing a significant level of depressive symptoms.
Anxiety | Change from baseline to 12-month post-intervention
  The State Anxiety Scale for Children (SAS-C), which is a 20-item subscale of the State-Trait Anxiety Scales Inventory for Children will be used to measure children's levels of anxiety. It is rated on a three-point Likert scale from 1 to 3 to indicate the degree to which an individual is experiencing a particular feeling at present.
Self-esteem | Change from baseline to 12-month post-intervention
  The Chinese version of the Rosenberg self-esteem scale (RSES) will be used to assess children's level of self-esteem. The scale contains 10 items, which are rated on a 4-point Likert scale with score 1 to 4 (1= strongly disagree, 2= disagree, 3= agree, 4 = strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.
Quality of life | Change from the baseline to 12-month post-intervention
  The Chinese version of the Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0) will be used to assess children's health-related quality of life. The scale consists of 23 items which are categorised into four dimensions, namely physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). All items are rated on a 5-point Likert scale from 0 (never) to 4 (almost always). Higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No